CLINICAL TRIAL: NCT01767285
Title: A Randomized Controlled Trial of Immediate Postpartum Etonogestrel Implant Versus Six-week Postpartum Etonogestrel Implant: A Pilot Study
Brief Title: Immediate vs. Delayed Postpartum Etonogestrel Implant
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00030001
Record Dates: First submitted 2013-01-07; First posted 2013-01-14 (Estimated); Results first posted 2016-12-19 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-01

CONDITIONS: Continuation Rate of Contraceptive Implant
Keywords: Etonogestrel Implant; Implanon; Nexplanon; Long Acting Reversible Contraception
MeSH Terms: interventions — etonogestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate Postpartum Etonogestrel Implant (Experimental): Etonogestrel implant placed in the hospital after delivery, before discharge home.
  Interventions: Drug: Etonogestrel implant
- Delayed postpartum etonogestrel implant (Active Comparator): These subjects will have the etonogestrel implant placed at the 6 week postpartum visit.
  Interventions: Drug: Etonogestrel implant

INTERVENTIONS:
Drug: Etonogestrel implant — This will be placed in subjects in both arms. Those in Arm 1 will receive the implant in the hospital postpartum. Those in Arm 2 will receive the implant at the 6 week postpartum visit.
  Other Names: Implanon; Nexplanon

SUMMARY:
The investigators are examining if there is a difference in continuation rates of the etonogestrel contraceptive implant between women who have the device placed immediately after delivery, before leaving the hospital, and women who have the device placed at the routine 6-week postpartum visit. There will be 60 subjects total, randomized in a 1:1 ratio, for 30 in each group. All participants will follow-up at the same postpartum clinic 6 weeks after delivery. They will then be contacted at 3, 6, and 12 months postpartum and asked to complete a brief survey. The investigators hypothesize that continuation rates of Implanon will be higher in the immediate postpartum placement arm than in the delayed placement arm.

ELIGIBILITY:
Inclusion Criteria:

1)Age 12-40 years 2)Must deliver at Duke Hospital 3)Must have a working telephone number 4)No contraindications to receiving this method of contraception, which include: known or suspected pregnancy, active liver disease or hepatic tumor, current or past history of thrombosis or thromboembolic disorder, undiagnosed abnormal genital bleeding, known or suspected breast cancer or history of breast cancer, hypersensitivity to any of the components of the device.

-

Exclusion Criteria:

1. Not meeting inclusion criteria
2. Use of chronic medical therapy that has an adverse interaction with etonogestrel. Medications that will be cause for exclusion from the study include:

1. Non-nucleoside reverse transcriptase inhibitors 2. ritonavir-boosted protease inhibitors 3. Certain anticonvulsants - phenytoin, carbamazepine, barbiturates, primidone, topiramate, oxcarbazepine 4. Rifampin 5. St. John's Wort

-

Ages: 12 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2013-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Morse, MD, Principal Investigator — Duke Hospital Department of Obstetrics and Gynecology
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Finer LB, Henshaw SK. Disparities in rates of unintended pregnancy in the United States, 1994 and 2001. Perspect Sex Reprod Health. 2006 Jun;38(2):90-6. doi: 10.1363/psrh.38.090.06. PMID 16772190
- [Background] Espey E, Ogburn T. Long-acting reversible contraceptives: intrauterine devices and the contraceptive implant. Obstet Gynecol. 2011 Mar;117(3):705-719. doi: 10.1097/AOG.0b013e31820ce2f0. PMID 21343774
- [Background] Guazzelli CA, de Queiroz FT, Barbieri M, Torloni MR, de Araujo FF. Etonogestrel implant in postpartum adolescents: bleeding pattern, efficacy and discontinuation rate. Contraception. 2010 Sep;82(3):256-9. doi: 10.1016/j.contraception.2010.02.010. Epub 2010 Mar 29. PMID 20705154
- [Background] Lewis LN, Doherty DA, Hickey M, Skinner SR. Implanon as a contraceptive choice for teenage mothers: a comparison of contraceptive choices, acceptability and repeat pregnancy. Contraception. 2010 May;81(5):421-6. doi: 10.1016/j.contraception.2009.12.006. Epub 2010 Jan 15. PMID 20399949
- [Background] Croxatto HB, Urbancsek J, Massai R, Coelingh Bennink H, van Beek A. A multicentre efficacy and safety study of the single contraceptive implant Implanon. Implanon Study Group. Hum Reprod. 1999 Apr;14(4):976-81. doi: 10.1093/humrep/14.4.976. PMID 10221230
- [Background] Funk S, Miller MM, Mishell DR Jr, Archer DF, Poindexter A, Schmidt J, Zampaglione E; Implanon US Study Group. Safety and efficacy of Implanon, a single-rod implantable contraceptive containing etonogestrel. Contraception. 2005 May;71(5):319-26. doi: 10.1016/j.contraception.2004.11.007. PMID 15854630
- [Background] Brito MB, Ferriani RA, Quintana SM, Yazlle ME, Silva de Sa MF, Vieira CS. Safety of the etonogestrel-releasing implant during the immediate postpartum period: a pilot study. Contraception. 2009 Dec;80(6):519-26. doi: 10.1016/j.contraception.2009.05.124. Epub 2009 Jul 10. PMID 19913145
- [Derived] Sothornwit J, Kaewrudee S, Lumbiganon P, Pattanittum P, Averbach SH. Immediate versus delayed postpartum insertion of contraceptive implant and IUD for contraception. Cochrane Database Syst Rev. 2022 Oct 27;10(10):CD011913. doi: 10.1002/14651858.CD011913.pub3. PMID 36302159

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 60 participants signed consent. 1 participant was a screen failure. 59 participants were randomized.
Period: Overall Study
Arm/Group | Immediate Postpartum Etonogestrel Implant | Delayed Postpartum Etonogestrel Implant
Started | 29 | 30
Completed | 22 | 24
Not Completed | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Postpartum Etonogestrel Implant | Delayed Postpartum Etonogestrel Implant | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 30 | 59
  >=65 years | 0 | 0 | 0
Gender [Count of Participants; unit: Participants]
  Female | 29 | 30 | 59
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 29 | 58

OUTCOME MEASURES:

1. Primary Outcome: Continuation Rate
Description: To identify a difference in continuation rates of Implanon® between women who have the device placed immediately postpartum and women who have the device placed at the 6-week postpartum visit.
Time Frame: 1 year
Population: Participants who completed the 1 year phone visit were included in analysis.
Measure: Number; unit: participants
Arm/Group | Immediate Postpartum Etonogestrel Implant | Delayed Postpartum Etonogestrel Implant
Number analyzed (Participants) | 22 | 21
participants | 20 | 18

2. Secondary Outcome: Rate of Intercourse
Description: To identify differences in the rates of intercourse prior to the 6-week postpartum visit.
Time Frame: 6 weeks
Population: Participants who completed the 6 week assessment.
Measure: Number; unit: participants
Arm/Group | Immediate Postpartum Etonogestrel Implant | Delayed Postpartum Etonogestrel Implant
Number analyzed (Participants) | 26 | 28
participants | 8 | 14

3. Secondary Outcome: Continuation Rate
Description: To identify a difference in continuation rates of Implanon® at one year between women who have the device placed immediately postpartum and women who have the device placed at the 6-week postpartum visit.
Time Frame: 6 months
Population: Participants who completed the 6 month assessment.
Measure: Number; unit: participants
Arm/Group | Immediate Postpartum Etonogestrel Implant | Delayed Postpartum Etonogestrel Implant
Number analyzed (Participants) | 27 | 28
participants | 27 | 21

4. Other Pre Specified Outcome: Continuation of Breastfeeding
Description: To identify differences in continuation of breast-feeding at 6 months between women who have immediate versus delayed (6 weeks) postpartum Implanon® placement.
Time Frame: 6 months
Population: Participants who completed the 6 month assessment.
Measure: Number; unit: participants
Arm/Group | Immediate Postpartum Etonogestrel Implant | Delayed Postpartum Etonogestrel Implant
Number analyzed (Participants) | 27 | 28
participants | 6 | 5

5. Other Pre Specified Outcome: Pregnancy Rate
Description: To identify differences pregnancy rates between women who have immediate versus delayed (6 weeks) postpartum Implanon® placement.
Time Frame: 12 months
Population: all participants who completed the 12 month follow up visit
Measure: Number; unit: participants
Arm/Group | Immediate Postpartum Etonogestrel Implant | Delayed Postpartum Etonogestrel Implant
Number analyzed (Participants) | 22 | 24
participants | 0 | 1

6. Other Pre Specified Outcome: Patient Satisfaction
Description: To identify differences in satisfaction with birth control method between women who have immediate versus delayed (6 weeks) postpartum Implanon® placement.
Time Frame: 12 months
Population: Participants who completed the 12 month patient satisfaction assessment.
Measure: Number; unit: participants
Arm/Group | Immediate Postpartum Etonogestrel Implant | Delayed Postpartum Etonogestrel Implant
Number analyzed (Participants) | 22 | 21
participants | 15 | 13

ADVERSE EVENTS:
Arm/Group | Immediate Postpartum Etonogestrel Implant | Delayed Postpartum Etonogestrel Implant
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 0/29 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes